CLINICAL TRIAL: NCT06595693
Title: Measurement and Prediction of Tilt and Decentration of the Clareon Intraocular Lens and Evaluation of It's Effect of Visual Acuity
Brief Title: Tilt Prediction of Clareon Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: JKU-Ophthalmology-001
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cataract
Keywords: Intraocular Lens; tilt; cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Misalignment of intraocular lenses can cause severe loss of visual quality. Different types of misalignments are known. Tilt, one type of intraocular lens misalignment is thought to play a negative role for the optical performance in eyes with intraocular designs, especially, if they have aspheric, toric, or multifocal optics. Various methods to measure intraocular lens misalignments have been described. The most recently developed method for tilt quantification is the use of optical coherence tomography. This method has several advantages compared to the previous methods: optical coherence tomography based devices are available in most clinics, the resolution of modern optical coherence tomography devices is high, and the measurements are reproducible.

DETAILED DESCRIPTION:
During cataract surgery an artificial intraocular lens is implanted in the eye to replace the lens and to correct the refraction for distance vision. Misalignment of intraocular lenses can cause severe loss of visual quality. Different types of misalignments are known. Tilt, one type of intraocular lens misalignment is thought to play a negative role for the optical performance in eyes with intraocular lens designs, especially, if they have aspheric, toric, or multifocal optics. For example, in the case of aspheric intraocular lenses, it appears that even slight amount of tilt may result not only in the loss of the effect of reducing spherical aberrations but in more severe cases even a worsening of the optical quality compared to spherical intraocular lenses. In the case of toric intraocular lenses, tilt introduces higher order aberrations potentially mimicking astigmatism. In the case of multifocal intraocular lenses, tilt increases higher order aberrations, which leads to decreased visual quality.

Various methods to measure intraocular lens misalignments have been described. Studies assessing the intraocular lens position have used subjective grading methods at the slit lamp examination or a Scheimpflug camera to assess intraocular lens decentration and tilt. The subjective grading at the slitlamp may display considerable variability between examiners. This method is more qualitative than quantitative and does not allow fine resolution when reporting intraocular lens tilt. The fact that the patient has no standardized target to focus on makes the method even less reliable. Scanning methods such as Scheimpflug photos require a very well dilated pupil exceeding 6mm to assess the intraocular lens position. Additionally, it can be difficult to identify the anatomical structures of the eye that need to be used as points of reference. Scheimpflug camera images have been used for assessing intraocular lens tilt previously, but erroneous results, often due to corneal magnification, have diminished their widespread use. Another possibility to assess tilt is the use of Purkinje reflexes. The light reflections of Purkinje images at ocular surfaces to evaluate ocular alignment have recently been utilized. Since light is reflected at all interfaces of media with a difference in refractive index, these reflections, called Purkinje images, can be used to assess tilt and decentration of intraocular lenses. Two different clinically applicable Purkinjemeter system provide the measurement of intraocular decentration and tilt. The main problem with Purkinje meters is accessibility, as there are only a few prototypes available worldwide.

The most recently developed method for tilt quantification is the use of optical coherence tomography. This method has several advantages compared to the previous methods: optical coherence tomography based devices are available in most clinics, the resolution of modern optical coherence tomography devices is high, and the measurements are reproducible.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract surgery in both eyes (bilateral inclusion only)
* Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visits
* Ability to consent to the participation in the study;
* Signed informed consent

Exclusion Criteria:

* Combined surgery (cataract plus glaucoma/vitreoretinal/corneal surgery)
* Best corrected distance visual acuity below 0.1 Snellen before surgery
* Pathologies that could have an influence on the post-operative tilt, such as pseudoexfoliation syndrome or previous ophthalmic trauma, or other reasons for phakodonesis
* Previous ophthalmic surgery that could have an influence on post-operative tilt, such as pars plana vitrectomy
* Pregnancy (pregnancy test will be taken preoperatively)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with planned cataract surgery of both eyes
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
post operative intraocular lens tilt in degrees measured between three different OCT based devices | 8 weeks post cataract surgery
  amount of tilt of intraocular lens post cataract surgery

SECONDARY OUTCOMES:
orientation of post operative tilt in degrees measured between three different OCT based devices | 8 weeks post cataract surgery
  Orientation of post operative tilt in degrees measured with three different optical coherence tomography devices.
decentration of intraocular lens in millimeter measured between three different OCT based devices | 8 weeks post cataract surgery
  Decentration of intraocular lens in millimeter is being determined with three different optical coherence tomography devices and compared to a Scheimpflug camera.
distance corrected visual acuity in logMAR | 8 weeks post cataract surgery
  Distance corrected visual acuity in logMAR will be determined by Best Corrected Visual Acuity

OTHER OUTCOMES:
visual acuity in logMAR in a subgroup of eyes | 8 weeks post cataract surgery
  visual acuity in logMAR in a subgroup of eyes with tilt greater than 5 degrees or less than 5 degrees determined by Best Corrected Visual Acuity

CONTACTS AND LOCATIONS:
Overall Officials: Nino Hirnschall, MD, Principal Investigator — JKU Linz
Locations (1):
- Department for Ophthalmology and Optometry, Kepler University Hospital GmbH, Johannes Kepler University Linz, Altenberger Strasse 69, 4040 Linz, Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waser K, Strassmair K, Pomberger L, Khalil H, Laubichler P, Bolz M, Hirnschall N. Capsular Bag Performance of a Novel Hydrophobic Single-Piece Intraocular Lens. Ophthalmol Ther. 2025 Feb;14(2):295-308. doi: 10.1007/s40123-024-01075-x. Epub 2024 Dec 12. PMID 39666249